CLINICAL TRIAL: NCT04856514
Title: Effectiveness of a Telehealth Group for Improving Peer Relationships for Adolescents With Neurofibromatosis Type 1
Brief Title: Open Trial of Telehealth Group for Improving Peer Relationships (PEERS) in NF1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: NF Midwest (Unknown)
Responsible Party: Principal Investigator, Bonita P Klein-Tasman, Professor, University of Wisconsin, Milwaukee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-039-UWM-a
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Neurofibromatosis 1; Social Skills
MeSH Terms: conditions — Neurofibromatosis 1; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Participation in 16 week telehealth administration of the PEERS protocol for teens (parallel teen and parent/caregiver groups)
  Interventions: Behavioral: PEERS

INTERVENTIONS:
Behavioral: PEERS — 16 week telehealth intervention; parallel teen and parent/caregiver groups; 90 minutes each week.

SUMMARY:
This is an open trial of the UCLA PEERS protocol delivered via Telehealth with teens with neurofibromatosis type 1 whose parents report that they have difficulty making and keeping friends.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of neurofibromatosis type 1
* Age 12-17
* Main language spoken in the home is English
* Reliable internet access
* Current functional impairment in peer relationships
* Teen is interested and motivated to participate

Exclusion Criteria:

* Main language spoken in the home is not English
* Cognitive or developmental delays that affect reading comprehension or understanding of treatment material
* Significant behavioral concerns
* Other comorbid medical conditions
* Major surgery in past 6 months
* Prior social skills group treatment within past 6 months
* Prior participation in PEERS

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) | within four weeks of PEERS completion
  Parental report of social skills (SSIS-SEL Total Score; Mean 100, SD 15; Higher scores mean stronger social functioning
Test of Adolescent Social SKills (TASSK: Laugeson & Frankel, 2010) | within four weeks of PEERS completion
  Questionnaire completed by teen participants; measures knowledge of the PEERS intervention concepts (raw total score; higher score means stronger functioning)

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS; Constantino, 2005) | within four weeks of PEERS completion
  Questionnaire completed by caregivers on social function and autism symptoms (SRS Total Score; Mean 50, SD 10; higher scores mean greater difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Glad, M.S., Study Director — University of Wisconsin, Milwaukee
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon request to qualitied investigators.
Supporting Information: Study Protocol, ICF
Time Frame: Available following publication of the research findings
Access Criteria: Contact the PI (bklein@uwm.edu)